CLINICAL TRIAL: NCT00092638
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Evaluate Efficacy, Safety, and Tolerability of Ezetimibe 10 mg or Placebo Added to Existing Atorvastatin 10 mg or 20 mg in Attaining Low-Density Lipoprotein Cholesterol Target Levels in Patients With Hypercholesterolemia and Coronary Heart Disease.
Brief Title: An Investigational Drug Study in Patients With Elevated Cholesterol and Coronary Heart Disease (0653-804)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0653-804; 2004_042
Record Dates: First submitted 2004-09-23; First posted 2004-09-27 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia; Coronary Disease
Keywords: Elevated Cholesterol
MeSH Terms: conditions — Hypercholesterolemia; Coronary Disease | interventions — Ezetimibe

INTERVENTIONS:
Drug: MK0653, ezetimibe
Drug: Comparator: ezetimibe, placebo

SUMMARY:
The purpose of this study is to investigate additional cholesterol lowering effects in patients with coronary heart disease by giving an investigational drug with a patient's current approved cholesterol lowering medication.

DETAILED DESCRIPTION:
The duration of treatment is 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with elevated cholesterol and coronary heart disease

Exclusion Criteria:

* Patients whose cholesterol levels measure within acceptable ranges as specified by the study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2003-05; Primary Completion 2004-07 (Actual); Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
Percentage of patients reaching their target LDL-C goal of </= 2.60 mmol/L, after 6 weeks of treatment.

SECONDARY OUTCOMES:
Safety and tolerability.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Cruz-Fernandez JM, Bedarida GV, Adgey J, Allen C, Johnson-Levonas AO, Massaad R. Efficacy and safety of ezetimibe co-administered with ongoing atorvastatin therapy in achieving low-density lipoprotein goal in patients with hypercholesterolemia and coronary heart disease. Int J Clin Pract. 2005 Jun;59(6):619-27. doi: 10.1111/j.1368-5031.2005.00565.x. PMID 15924587